CLINICAL TRIAL: NCT03678961
Title: Influence of Lower Extremity Positioning During Anterior-approach Ultrasound-guided Sciatic Nerve Block: Depth and Visibility
Brief Title: The Effect of Leg Position on the Sciatic Nerve on Sonogram
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hajung Kim, Clinical Instructor, Asan Medical Center
Other Study IDs: 2018-0970
Record Dates: First submitted 2018-08-17; First posted 2018-09-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Sciatic Nerve Block

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group N: Neutral position
- Group E: External rotation of leg by 45 degrees
  Interventions: Behavioral: external rotation of leg
- Group EF45: External rotation of leg by 45 degrees, hip flexion by 45 degrees, and knee flexion by 45 degrees
  Interventions: Behavioral: external rotation of leg; Behavioral: hip flexion and knee flexion
- Group EF15: External rotation of leg by 45 degrees, hip flexion by 15 degrees, and knee flexion by 15 degrees
  Interventions: Behavioral: external rotation of leg; Behavioral: hip flexion and knee flexion

INTERVENTIONS:
Behavioral: external rotation of leg — external rotation of leg by 45 degrees
  Groups: Group E; Group EF15; Group EF45
Behavioral: hip flexion and knee flexion — hip flexion by 15/45 degrees and knee flexion by 15/45 degrees
  Groups: Group EF15; Group EF45

SUMMARY:
Little is known about which posture of lower extremity makes it easier to access to the sciatic nerve. In this study, the investigators aimed to identify the most appropriate positioning of the lower extremity during anterior-approach ultrasound-guided sciatic nerve block.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS 1-3
* patients undergoing knee surgery requiring peripheral nerve block

Exclusion Criteria:

* patients who refuse to participate in the study
* BMI > 40 kg/m2
* patients who have congenital abnormality on leg
* patients who have surgery or trauma on hip/knee
* patients who cannot move freely due to the contracture
* patients who are judged ineligible by the medical staff to participate in the study for other reasons

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing knee surgery requiring peripheral nerve block
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Visibility of sciatic nerve | during 10 minutes of anesthesia induction
  Visibility of sciatic nerve at each position assessed using a scoring system (0, no nerve identified; 1, nerve identified with a high probability; 2, nerve identified, but most of it not visible; 3, nerve identified, more than 50% of its borders can be precisely distinguished from surrounding structures; 4, nerve completely visible, but fascicles poorly defined; 5, nerve completely visible and multiple fascicles identifiable.)

SECONDARY OUTCOMES:
Depth of sciatic nerve | during 10 minutes of anesthesia induction
  Distance from skin to sciatic nerve at each position

CONTACTS AND LOCATIONS:
Overall Officials: Won Uk Koh, M.D., Ph.D., Principal Investigator — University of Ulsan, College of Medicine, Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea